CLINICAL TRIAL: NCT04268849
Title: A Randomized, Placebo-controlled Comparator Trial of IV vs Oral Iron Treatment of Iron Deficiency Anemia in the Post-Operative Bariatric Surgical Patient
Brief Title: Trial of IV vs Oral Iron Treatment of Iron Deficiency Anemia in the Post-Operative Bariatric Surgical Patient
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Auerbach Hematology Oncology Associates P C (Other)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Auerbach MD, Principal Investigator, Auerbach Hematology Oncology Associates P C
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BariatricsProtocol100719
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Iron Deficiency Anemia
Keywords: Bariatric Surgery; Roux-en-Y gastric bypass (RYGB); Vertical Sleeve Gastrectomy (VSG)
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferrosoferric Oxide; Sodium Chloride; Iron-Dextran Complex; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Double blind, double dummy of oral versus intravenous iron for iron deficiency patients after bariatric surgery. All subjects will get either oral iron and intravenous saline, or oral vitamin C and intravenous iron.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will wear sleep masks to blind intravenous intervention
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral Iron (Active Comparator): The subject will receive one IV infusion of ferumoxytol administered as 1020 mg over 30 minutes or an equivalent volume of normal saline. At the time of the infusion, the patient will also be given an opaque bottle, containing either vitamin C tablets or ferrous sulfate 325 mg.
  Interventions: Drug: Ferumoxytol; Drug: Saline; Drug: Ferrous sulfate tablets; Drug: Vitamin C
- IV Iron (Active Comparator): The subject will receive one IV infusion of ferumoxytol administered as 1020 mg over 30 minutes or an equivalent volume of normal saline. At the time of the infusion, the patient will also be given an opaque bottle, containing either vitamin C tablets or ferrous sulfate 325 mg.
  Interventions: Drug: Ferumoxytol; Drug: Saline; Drug: Ferrous sulfate tablets; Drug: Vitamin C

INTERVENTIONS:
Drug: Ferumoxytol — Ferumoxytol (30 mg/mL) intravenous injection in single use vials.
Drug: Saline — Placebo for Ferumoxytol
Drug: Ferrous sulfate tablets — ferrous sulfate tablets containing 60 mg elemental iron
Drug: Vitamin C — Placebo: Vitamin C, 250 mg, given in the same bottle as the oral iron

SUMMARY:
Given the limited long-term effectiveness of traditional weight loss methods, bariatric surgery is increasingly becoming the preferred option for sustained weight loss. With the ascendancy of the laparoscopic approach, the two most common procedures are the Roux-en-Y gastric bypass (RYGB) and the vertical sleeve gastrectomy (VSG).

Because bariatric surgery decreases nutrient intake through restriction, malabsorption, or both, and given that obese patients are often malnourished even before surgery, postoperative micronutrient deficiency, particularly of iron, can be a serious complication and difficult to treat. Iron deficiency anemia has been reported to be as high as 49% in the post-bariatric surgical patient.

The current standard for correcting iron deficiency anemia in the post-operative bariatric surgical patient is oral iron supplements. However, oral iron therapy is known for its caustic effects on the gastric mucosa causing gastric irritation, nausea, epigastric discomfort and constipation. These debilitating symptoms lead to poor adherence and lower long and short-term efficacy. Furthermore, iron absorption from oral iron supplements when taken with food in patients with low iron stores ranges from 2 to 13% and without food 5 to 28%. An alternative and more effective method of iron replenishment is the use of intravenous iron. A litany of published trials, without contradiction, show marked superiority of intravenous iron in improving hemoglobin concentrations and iron parameters when compared to historical controls. Nonetheless, the current recommendations of the American Society of Metabolic and Bariatric Surgery nutritional guidelines, state that oral iron supplementation for IDA is the recommended first line of treatment. Studies are lacking that compare the efficacy of oral versus intravenous (IV) iron therapy for the treatment of IDA in the post-bariatric surgical patient.

The aim of our study is to compare two accepted treatments for iron deficiency anemia (oral ferrous sulfate and intravenous ferumoxytol) for efficacy and speed of response in the treatment of IDA in the post-operative bariatric surgical patient. In this study, 104 bariatric surgical post-operative patients will be randomly assigned 52 each to oral or 52 to a single dose IV iron treatment using double-blind procedures.

The primary outcome will be determined at 6 weeks of treatment with a follow-up at 12 months after treatment. Non-responders at 6 weeks after treatment may, if they qualify (based on inclusion/exclusion criteria), have an open-label IV iron treatment and will be followed with the same evaluations used after the first IV iron treatments.

ELIGIBILITY:
Inclusion criteria:

1. Aged ≥ 18 years
2. Patients who have undergone a Roux-en Y Gastric Bypass or Vertical Sleeve Gastrectomy and are at least 3 months or more out from surgery.
3. Iron deficiency anemia defined as iron deficient with either ferritin<30 mcg/l, TSAT<20%, or anemia with Hgb<13 g/dL for both males and females.
4. Willingness to participate and signing the informed consent form.

Exclusion criteria:

1. Iron overload or disturbances in utilization of iron (e.g. hemochromatosis and hemosiderosis)
2. Decompensated liver cirrhosis or active hepatitis (ALAT > 3 times upper limit of normal)
3. Serum ferritin > 400 ng/mL or transferrin saturation >40 %
4. Active acute or chronic infections (assessed by clinical judgment that may be indicated by White Blood Cells (WBC) and C-Reactive Protein (CRP) when these are available)
5. Rheumatoid arthritis with symptoms or signs of active inflammation
6. Pregnant and nursing women
7. History of multiple allergies (two or more)
8. Known hypersensitivity to ferumoxytol or oral iron or any excipients in the drug products
9. Previous IV iron treatment for IDA
10. Other iron treatment or blood transfusion within 4 weeks prior to the screening or treatment visit
11. Planned elective surgery during the study
12. Any other medical condition that, in the opinion of Investigator, may cause the subject to be unsuitable for the completion of the study or place the subject at potential risk from being in the study, e.g. a malignancy, uncontrolled hypertension, unstable ischemic heart disease, or uncontrolled diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Global Impression - improvement scale (CGI-2) score at 6 weeks after treatment begins. | 6 weeks
  The CGI-2 is a measure of treatment response and the efficacy of the treatment based on a 1 to 7 scale where 1 is "very much better" and 7 "very much worse"
Change in hemoglobin concentration | 6 weeks

SECONDARY OUTCOMES:
Change in ferritin > 20% | 6 weeks
Change in Transferrin saturation (TSAT) >19% | 6 weeks
Quality of Life by visual linear analog scale (LASA) | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Auerbach Hematology and Oncology, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No